CLINICAL TRIAL: NCT05195242
Title: The Effect of Dexamethasone 12 mg vs 6 mg on Thromboembolic Events in Patients With Critical COVID-19 - a Post-hoc Analysis of the Blinded, Randomized COVID STEROID 2 Trial
Brief Title: The Effect of Dexamethasone 12 mg vs 6 mg on Thromboembolic Events in Patients With Critical COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Scandinavian Critical Care Trials Group (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Centre for Research in Intensive Care (CRIC) (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other); Linkoeping University (Other Government); Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Sandra Jonmarker, MD, Consultant in Intensive Care and Anaesthesiology, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Thromboembolism COVIDSTEROID2
Record Dates: First submitted 2022-01-13; First posted 2022-01-18 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Thrombosis Embolism; Bleeding
MeSH Terms: conditions — COVID-19; Embolism and Thrombosis; Hemorrhage | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone 12 mg (Experimental): Intravenous bolus injection of dexamethasone 12 mg once daily in addition to standard care for up to 10 days. We will allow the use of betamethasone 12 mg at sites, where dexamethasone is not available.
  Interventions: Drug: Dexamethasone
- Dexamethasone 6 mg (Active Comparator): Intravenous bolus injection of dexamethasone 6 mg once daily in addition to standard care for up to 10 days. We will allow the use of betamethasone 6 mg at sites, where dexamethasone is not available.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — ATC code H02AB02
  Other Names: Dexavit

SUMMARY:
Thromboembolisms (TEs) in patients with critical COVID-19 has been reported to be three times higher than for other critically ill patients. Immunothrombosis has been proposed as a plausible mechanism for COVID-19 coagulopathy. Corticosteroids improve survival in patients with critical COVID-19, and likely even more so with a higher dose. However, the evidence regarding the impact on the incidence of thromboembolic and bleeding events are currently uncharted. The aim of this study is to investigate if there is a difference in the incidence of thromboembolic events during ICU stay in patients with critical COVID-19 when treated with 12 mg dexamethasone compared to 6 mg dexamethasone.

ELIGIBILITY:
All patients were recruited from the CS2-trial with following inclusion/exclusion criteria:

Inclusion Criteria:

* confirmed SARS-CoV-2 AND
* requiring at least 10l/min of O2 supplementation, non-invasive mechanical ventilation for hypoxia or invasive mechanical AND

Exclusion Criteria:

* if previously randomised to the CS2 trial
* if they had received corticosteroids for COVID-19 during ≥5 consecutive days or use corticosteroids in doses >6 mg dexamethasone for an indication other than COVID-19.
* active tuberculosis
* hypersensitivity to dexa-/betamethasone
* active fungal infection
* fertile woman ≤60 years of age with a positive U-HCG/P-HCG test
* informed consent not obtainable

For the inclusion in this post-hoc analyses there is additional criteria:

Inclusion Criteria:

- randomised in the ICU

Exclusion Criteria:

* established thromboembolism at randomisation
* established major bleeding at randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients discharged alive from the ICU without thromboembolic events | During ICU-stay
  Number of patients discharged alive from the ICU without thromboembolic events defined as pulmonary embolism, deep venous thrombosis, ischemic stroke, myocardial infarction, transient ischemic attack, other thromboembolic events

SECONDARY OUTCOMES:
The cumulative proportion of thromboembolic events | During ICU-stay
  The incidence of thromboembolic events defined as pulmonary embolism, deep venous thrombosis, ischemic stroke, myocardial infarction, transient ischemic attack, other thromboembolic events
The cumulative proportion of bleeding events | During ICU-stay
  The cumulative proportion of bleeding events defined as any type of bleeding
The cumulative proportion of major bleeding events | During ICU-stay
  The cumulative proportion of major bleeding event (defined as bleeding requiring transfusion of at least 2 units of Red Blood Cells (RBC) and/or intracranial bleeding and/or bleeding resulting in need for major therapeutic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rebecka Rubenson Wahlin, MD. PhD, Study Director — Karolinska Institutet Södersjukhuset; Maria Cronhjort, MD PhD, Study Chair — Karolinska Institutet Södersjukhuset
Locations (1):
- Södersjukhuset, Stockholm, Stockholm County, Sweden